CLINICAL TRIAL: NCT04381819
Title: Norwegian SARS-CoV-2 Study - Virological, Clinical and Immunological Characterisation of Inpatients During the COVID-19 Outbreak: A Prospective Cohort Study
Brief Title: Norwegian SARS-CoV-2 Study - Virological, Clinical and Immunological Characterisation of COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: University Hospital, Akershus (Other); Vestre Viken Hospital Trust (Other); Ostfold Hospital Trust (Other); Haukeland University Hospital (Other); University Hospital of North Norway (Other); St. Olavs Hospital (Other)
Responsible Party: Principal Investigator, Jan Cato Holter, Project leader, medical doctor, PhD, Oslo University Hospital
Other Study IDs: 20-04072
Record Dates: First submitted 2020-05-04; First posted 2020-05-11 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: SARS Virus; Severe Acute Respiratory Syndrome
MeSH Terms: conditions — Severe Acute Respiratory Syndrome | interventions — COVID-19 Nucleic Acid Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Respiratory secretions, blood, urine, stool, cerebrospinal fluid
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: SARS-CoV-2 PCR — SARS-CoV-2 E gene

SUMMARY:
Oslo University Hospital has initiated an observational study on hospitalised patients with confirmed COVID-19, the infection caused by Severe Acute Respiratory Syndrome Coronavirus type 2 (SARS-CoV-2).

DETAILED DESCRIPTION:
Infectious disease is the single biggest cause of death worldwide. New infectious agents, such as the SARS-CoV-2, require investigation to understand pathogen biology and pathogenesis in the host. In order to develop a mechanistic understanding of disease processes, such that risk factors for severe illness can be identified and treatments can be developed, it is necessary to understand pathogen characteristics associated with virulence, the replication dynamics and in-host evolution of the pathogen, the dynamics of the host response, the pharmacology of antimicrobial or host directed therapies, the transmission dynamics, and factors underlying individual susceptibility.

At Oslo University Hospital, an observational study on the newly discovered emerging SARS- CoV-2, the coronavirus that causes COVID-19 infection has started. The study has been approved by the Regional Ethics Committee, so that inclusion of confirmed COVID-19 cases admitted at the hospital can start immediately including the first patients needing hospitalisation. The plan is to include more hospitals in other parts of Norway, starting with inclusion of Akershus University Hospital, Vestre Viken Drammen Hospital and Østfold Hospital. The study is anticipated to provide much needed data on the course of the COVID-19 infection, as well as generating knowledge about the virus and its transmission.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed COVID-19 by screening of SARS-CoV-2 E-gene

Exclusion Criteria:

* Refusal of consent by patient or closest relative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Oslo University Hospital, Vestre Viken Drammen Hospital, Akershus University Hospital or Østfold Hospital Kalnes will be recruited consecutively after testing positive for SARS-CoV-2
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Death | From date of randomization until the date of death from any cause assessed up to 3 months.
  Fatal outcome from COVID-19
Recovery from COVID-19 | From date of randomization until the date of recovery from COVID-19 symptoms assessed up to 3 months.
  Resolved infection
Progression to ICU care or ventilation | 30 days
  Percentage of patients requiring intensive care admission or ventilation

SECONDARY OUTCOMES:
Clearance of SARS-CoV-2 from respiratory specimen | The number of calendar days from date of PCR positive test (counted as 1 day) in respiratory specimen until date of such test first become negative in the respiratory specimen assessed up to 3 months
  The change in(clearance of) viral RNA measured by polymerase chain reaction assay (PCR) test at days 1, 3, 8,14 and 90 days
Immune response to COVID-19 | From date of randomization until the date of clinical follow-up assessed up to 3 months.
  Cell-mediated and humoral immunity

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik G Müller, Professor, Study Director — University of Oslo; Susanne G Dudman, Professor, Study Chair — University of Oslo; Jan C Holter, PhD, Principal Investigator — Oslo University Hospital
Locations (7):
- Norway (7):
  - Vestre Viken Drammen Hospital, Drammen, Akershus
  - Haukeland University Hospital, Bergen
  - Østfold Hospital Trust, Fredrikstad
  - Akershus University Hospital, Lørenskog
  - Oslo University Hospital, Oslo
  - University Hospital North Norway, Tromsø
  - St Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Troseid M, Holter JC, Holm K, Vestad B, Sazonova T, Granerud BK, Dyrhol-Riise AM, Holten AR, Tonby K, Kildal AB, Heggelund L, Tveita A, Boe S, Muller KE, Jenum S, Hov JR, Ueland T; Norwegian SARS-CoV-2 study group. Gut microbiota composition during hospitalization is associated with 60-day mortality after severe COVID-19. Crit Care. 2023 Feb 23;27(1):69. doi: 10.1186/s13054-023-04356-2. PMID 36814280
- [Derived] Tveita A, Murphy SL, Holter JC, Kildal AB, Michelsen AE, Lerum TV, Kaarbo M, Heggelund L, Holten AR, Finbraten AK, Muller KE, Mathiessen A, Boe S, Fevang B, Granerud BK, Tonby K, Lind A, Dudman SG, Henriksen KN, Muller F, Skjonsberg OH, Troseid M, Barratt-Due A, Dyrhol-Riise AM, Aukrust P, Halvorsen B, Dahl TB, Ueland T; NOR-SOLIDARITY Consortium and the Norwegian SARS-CoV-2 Study Group Investigators. High Circulating Levels of the Homeostatic Chemokines CCL19 and CCL21 Predict Mortality and Disease Severity in COVID-19. J Infect Dis. 2022 Dec 13;226(12):2150-2160. doi: 10.1093/infdis/jiac313. PMID 35876699